CLINICAL TRIAL: NCT00783198
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Long-Term Safety of Ragweed (Ambrosia Artemisiifolia) Sublingual Tablet (SCH 39641) in Adult Subjects With a History of Ragweed-Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: Efficacy and Long-Term Safety of Ragweed (Ambrosia Artemisiifolia) Sublingual Tablet in Adults With a History of Ragweed-Induced Rhinoconjunctivitis With or Without Asthma (Study P05233)(COMPLETED)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05233; 2008-003863-38 (EudraCT Number); MK-3641-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis; Allergic, With Asthma; Conjunctivitis
MeSH Terms: conditions — Rhinitis; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SCH 39641 6 Amb a 1-U (Experimental): Participants receive Ambrosia artemisiifolia allergen extract (SCH 39641 6 Amb a 1-U) rapidly dissolving tablets, administered once daily sublingually for approximately 52 weeks
  Interventions: Biological: SCH 39641 6 Amb a 1-U
- SCH 39641 12 Amb a 1-U (Experimental): Participants receive Ambrosia artemisiifolia allergen extract (SCH 39641 12 Amb a 1-U) rapidly dissolving tablets, administered once daily sublingually for approximately 52 weeks
  Interventions: Biological: SCH 39641 12 Amb a 1-U
- Placebo (Placebo Comparator): Participants receive placebo matching ambrosia artemisiifolia allergen extract, rapidly dissolving tablets, administered once daily sublingually for approximately 52 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SCH 39641 6 Amb a 1-U — SCH 39641 6 Amb a 1-U sublingual tablets administered once daily
  Other Names: MK-3641
  Arms: SCH 39641 6 Amb a 1-U
Biological: SCH 39641 12 Amb a 1-U — SCH 39641 12 Amb a 1-U sublingual tablets administered once daily
  Other Names: MK-3641
  Arms: SCH 39641 12 Amb a 1-U
Biological: Placebo — matching placebo sublingual tablets administered once daily
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ragweed sublingual tablet (SCH 39641/MK-3641) compared with placebo in participants with ragweed-induced rhinoconjunctivitis over a one-year period. It is expected that ragweed allergic participants on one of the active arms of the trial will have decreased allergic rhinoconjunctivitis symptoms and require less allergy rescue medications during ragweed pollen season.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical history of significant ragweed-induced allergic rhinoconjunctivitis of at least 2 years duration, with or without asthma and have received treatment during the previous RS.
* Must have a positive skin prick test response to Ambrosia artemisiifolia at Screening Visit.
* Must be positive for specific immunoglobulin E (IgE) against Ambrosia artemisiifolia at Screening Visit.
* Must have an forced expiratory volume in 1 second (FEV1) of at least 70% of predicted at Screening Visit.
* Safety laboratory tests and vital signs conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor

Exclusion Criteria:

* Clinical history of symptomatic seasonal allergic rhinitis and/or asthma having received regular medication, due to another allergen during or potentially overlapping the RS.
* Clinical history of significant symptomatic perennial allergic rhinitis and/or asthma due to an allergen to which the participant is regularly exposed.
* Receipt of an immunosuppressive treatment within 3 months prior to the Screening Visit (except steroids for allergic and asthma symptoms).
* Clinical history of severe asthma.
* Asthma requiring medium or high dose inhaled corticosteroids.
* History of anaphylaxis with cardiorespiratory symptoms.
* History of chronic urticaria and angioedema.
* Clinical history of chronic sinusitis 2 years prior to the Screening Visit.
* Current severe atopic dermatitis.
* Breast-feeding, pregnant, or intending to become pregnant.
* Had previous treatment by immunotherapy with ragweed allergen or any other allergen 5 years prior to Screening Visit.
* History of allergy, hypersensitivity or intolerance to the ingredients of the investigational medicinal products (except for Ambrosia artemisiifolia), rescue medications, or self-injectable epinephrine.
* History of self-injectable epinephrine use.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 565 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

REFERENCES:
- [Derived] Christensen LH, Ipsen H, Nolte H, Maloney J, Nelson HS, Weber R, Lund K. Short ragweeds is highly cross-reactive with other ragweeds. Ann Allergy Asthma Immunol. 2015 Dec;115(6):490-495.e1. doi: 10.1016/j.anai.2015.09.016. Epub 2015 Oct 21. PMID 26507708
- [Derived] Kim H, Waserman S, Hebert J, Blaiss M, Nelson H, Creticos P, Kaur A, Maloney J, Li Z, Nolte H. Efficacy and safety of ragweed sublingual immunotherapy in Canadian patients with allergic rhinoconjunctivitis. Allergy Asthma Clin Immunol. 2014 Nov 10;10(1):55. doi: 10.1186/1710-1492-10-55. eCollection 2014. PMID 25788949
- [Derived] Nolte H, Amar N, Bernstein DI, Lanier BQ, Creticos P, Berman G, Kaur A, Hebert J, Maloney J. Safety and tolerability of a short ragweed sublingual immunotherapy tablet. Ann Allergy Asthma Immunol. 2014 Jul;113(1):93-100.e3. doi: 10.1016/j.anai.2014.04.018. Epub 2014 May 14. PMID 24836393
- [Derived] Nolte H, Hebert J, Berman G, Gawchik S, White M, Kaur A, Liu N, Lumry W, Maloney J. Randomized controlled trial of ragweed allergy immunotherapy tablet efficacy and safety in North American adults. Ann Allergy Asthma Immunol. 2013 Jun;110(6):450-456.e4. doi: 10.1016/j.anai.2013.03.013. Epub 2013 May 2. PMID 23706715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Started | 190 | 187 | 188
Completed | 133 | 144 | 146
Not Completed | 57 | 43 | 42
Not completed — Adverse Event | 15 | 19 | 3
Not completed — Lost to Follow-up | 11 | 1 | 7
Not completed — Withdrawal by Subject | 22 | 14 | 20
Not completed — Noncompliance with protocol | 7 | 7 | 10
Not completed — Did not meet protocol eligibility | 0 | 1 | 0
Not completed — Administrative | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo | Total
Number analyzed (Participants) | 190 | 187 | 188 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.00) | 34.9 (9.41) | 35.9 (9.13) | 35.4 (9.17)
Gender [Count of Participants; unit: Participants]
  Female | 84 | 109 | 93 | 286
  Male | 106 | 78 | 95 | 279

OUTCOME MEASURES:

1. Primary Outcome: Combined (Sum of) Rhinoconjunctivitis Daily Symptom Score (DSS) and Daily Medication Score (DMS) Averaged Over the Peak Ragweed Season (RS)
Description: The total combined score is a composite endpoint that combines the rhinoconjuntivitis DSS and the rhinoconjunctivitis DMS. The rhinoconjunctivitis DSS consisted of a total of 6 symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes and watery eyes) that were measured on a scale of 0 to 3 (0=no symptoms, 3=severe symptoms; score range: 0-18). Rhinoconjunctivitis DMS was based on participant use of specific study-provided rescue medicationwith different rescue medications being assigned different scores/dose unit. The maximum rhinoconjunctivitis DMS score was 36. The sum of the rhinoconjunctivitis DSS and DMS could range from 0 to 54, with a lower score indicating less rhinoconjuntivitis symptoms and medication use. Raw means for DSS+DMS were converted to adjusted means based on an analysis of variance (ANOVA) model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who took at least one dose of study medication and had at least one post-randomization efficacy measurement. A total of 5 participants at one site were excluded from all efficacy analyses due to Good Clinical Practice (GCP) issues.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 150 | 159 | 164
score on a scale | 6.70 (0.563) [-2.95 to -0.57] | 6.22 (0.543) [-3.41 to -1.07] | 8.46 (0.521) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0039, ANOVA; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-2.95 to -0.57] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0002, ANOVA; Mean Difference (Final Values) = -2.24, 95% CI 2-sided [-3.41 to -1.07] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

2. Secondary Outcome: Average Combined Rhinoconjunctivitis DSS and DMS Over the Entire RS
Description: The total combined score is a composite endpoint that combines the rhinoconjuntivitis DSS and the rhinoconjunctivitis DMS. The rhinoconjunctivitis DSS consisted of a total of 6 symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes and watery eyes) that were measured on a scale of 0 to 3 (0=no symptoms, 3=severe symptoms; score range: 0-18). Rhinoconjunctivitis DMS was based on participant use of specific study-provided rescue medicationwith different rescue medications being assigned different scores/dose unit. The maximum rhinoconjunctivitis DMS score was 36. The sum of the rhinoconjunctivitis DSS and DMS could range from 0 to 54, with a lower score indicating less rhinoconjuntivitis symptoms and medication use. Raw means for DSS+DMS were converted to adjusted means based on an ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: Approximately 5 weeks
Population: The FAS population consisted of all randomized participants who took at least one dose of study medication and had at least one post-randomization efficacy measurement. A total of 5 participants at one site were excluded from all efficacy analyses due to GCP issues.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 152 | 160 | 166
score on a scale | 5.92 (0.467) [-2.08 to -0.09] | 5.21 (0.450) [-2.78 to -0.82] | 7.01 (0.434) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0320, ANOVA; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-2.08 to -0.09] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0003, ANOVA; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-2.78 to -0.82] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

3. Secondary Outcome: Average Rhinoconjunctivitis DSS for the Peak RS
Description: The rhinoconjunctivitis DSS consisted of a total of 6 symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes and watery eyes) that were measured on a scale of 0 to 3 (0=no symptoms, 3=severe symptoms; score range: 0-18), with a lower score indicating less rhinoconjuntivitis symptoms. Raw means for DSS were converted to adjusted means based on an ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 150 | 159 | 164
score on a scale | 4.81 (0.362) [-1.54 to -0.01] | 4.65 (0.349) [-1.70 to -0.19] | 5.59 (0.335) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0472, ANOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.54 to -0.01] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0144, ANOVA; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.70 to -0.19] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

4. Secondary Outcome: Average Rhinoconjunctivitis DSS for the Entire RS
Description: as for outcome 3
Time Frame: Approximately 5 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 152 | 160 | 166
score on a scale | 4.41 (0.306) [-1.11 to 0.19] | 4.05 (0.295) [-1.46 to -0.18] | 4.87 (0.285) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.1686, ANOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.11 to 0.19] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0125, ANOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.46 to -0.18] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

5. Secondary Outcome: Average Rhinoconjunctivitis DMS for the Peak RS
Description: Rhinoconjunctivitis DMS was based on participant use of specific study-provided rescue medicationwith different rescue medications being assigned different scores/dose unit. The maximum rhinoconjunctivitis DMS score was 36, with a lower score indicating less rhinoconjuntivitis medication use. Raw means for DMS were converted to adjusted means based on an ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 150 | 159 | 164
score on a scale | 1.89 (0.314) [-1.65 to -0.32] | 1.57 (0.303) [-1.95 to -0.64] | 2.87 (0.291) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0039, ANOVA; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.65 to -0.32] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-1.95 to -0.64] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

ADVERSE EVENTS:
Time Frame: Up to 53 weeks
Description: A total of 5 participants (2 in the SCH 39641 6 Amb a 1-U group, 1 in the SCH 39641 12 Amb a 1-U group and 2 in the Placebo group) at one site were excluded from all safety analyses due to GCP issues. Adverse events are reported for the remaining participants.
Arm/Group | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Serious Adverse Events (participants affected / at risk) | 2/188 | 3/186 | 4/186
Other Adverse Events (participants affected / at risk) | 124/188 | 136/186 | 93/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 39641 6 Amb a 1-U (N=188) | SCH 39641 12 Amb a 1-U (N=186) | Placebo (N=186)
Pelvic mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 39641 6 Amb a 1-U (N=188) | SCH 39641 12 Amb a 1-U (N=186) | Placebo (N=186)
Ear pruritus (Ear and labyrinth disorders) | 30 (39) | 30 (33) | 4 (5)
Lip swelling (Gastrointestinal disorders) | 6 (10) | 14 (16) | 3 (4)
Nausea (Gastrointestinal disorders) | 6 (11) | 13 (16) | 2 (2)
Oral pruritus (Gastrointestinal disorders) | 36 (41) | 36 (44) | 6 (7)
Paraesthesia oral (Gastrointestinal disorders) | 14 (18) | 20 (28) | 4 (5)
Swollen tongue (Gastrointestinal disorders) | 22 (24) | 36 (51) | 6 (7)
Tongue pruritus (Gastrointestinal disorders) | 32 (41) | 27 (36) | 3 (3)
Nasopharyngitis (Infections and infestations) | 31 (41) | 27 (45) | 33 (42)
Sinusitis (Infections and infestations) | 9 (13) | 12 (14) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 22 (33) | 19 (26) | 28 (38)
Headache (Nervous system disorders) | 14 (19) | 20 (29) | 16 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 15 (16) | 5 (6)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (6) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 13 (15) | 9 (10)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 48 (73) | 55 (73) | 10 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (17) | 10 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.